CLINICAL TRIAL: NCT01518634
Title: Treatment of Multi-organ Bodily Distress Syndrome. A Double-blinded Placebo Controlled Trial of the Effects of Imipramine (Stress-3)
Brief Title: Imipramine Treatment for Patients With Multi-organ Bodily Distress Syndrome
Acronym: Stress-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-004294-87
Record Dates: First submitted 2012-01-13; First posted 2012-01-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-06

CONDITIONS: Somatisation Disorder; Somatoform Disorders
Keywords: Bodily Distress Syndrome; Medically unexplained symptoms; Functional somatic symptoms; Functional somatic syndromes; Treatment; Imipramine; Tricyclic antidepressant
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imipramine treatment (Experimental)
  Interventions: Drug: Imipramine treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imipramine treatment — Two-week of wash-out, one week of 10 mg study drug, 10 weeks of 25-75 mg study drug, four weeks of phasing-out and finaly two weeks after ther last dose of study drug to monito adverse events.
  Arms: Imipramine treatment
Drug: Placebo — Two-week of wash-out, one week of 10 mg study drug, 10 weeks of 25-75 mg study drug, four weeks of phasing-out and finaly two weeks after ther last dose of study drug to monito adverse events.
  Arms: Placebo

SUMMARY:
The aim of this study is to test the effect of the tricyclic antidepressant Imipramine in patients with longlasting health problems with no known medical explanation, defined as multi-organ Bodily distress syndrome (BDS). Pharmacological treatment of patients with BDS have never been tested, and Imipramine i low dosage (10-75 mg) has the potential of reducing both pain and other symptoms of bodily distress for patients with BDS. Control conditions are pill placebo. Study duration is 19 weeks for each of the 140 patients. End point is 13 weeks, i.e. after 10 weeks of 25-75 mg study drug.

DETAILED DESCRIPTION:
The aim of this study is to test the effect of Imipramine in patients with multi-organ Bodily distress syndrome (BDS). BDS is a unifying diagnosis that encompasses a group of closely related conditions such as somatization disorder, fibromyalgia, irritable bowel syndrome and chronic fatigue syndrome. The project consists of a double-blinded placebo controlled trial of treatment with the tricyclic antidepressant Imipramine in dosages of 25-75 mg. Primary outcome is patient-rated improvement measured by Clinical Global Improvement Scale (CGI-I). Secondary outcome is functional level (physical, mental and social) measured by the SF-36 Physical Component Summary (PCS). The study requires 140 participants and study duration is 19 weeks for each patient. End point is 13 weeks, i.e. after 10 weeks of 25-75 mg study drug.

ELIGIBILITY:
Inclusion Criteria:

1. First time refered patients fulfilling diagnostic criteria for BDS multi-organ type with symptoms for more than 3 of 4 symptom categories
2. Moderate or severe impact on daily life
3. Symptoms lasting for at least 2 years
4. Age 20-50 years
5. Born in Denmark or have Danish parents. The patient understands, speaks, writes and read Danish.

Exclusion Criteria:

1. Presence og other physical of psychiatric condition, if the symptoms of this condition can not clearly be separated from symptoms of BDS
2. Current moderate or severe depression, patients in continuous antidepressant treatment because of moderate or severe depression, and patients with other severe psychiatric disorder that demands treatment, or if the patient is suicidal.
3. A lifetime-diagnosis of psychoses, mania or depression with psychotic symptoms (ICD-10: F20-29, F30-31, F32.3, F33.3)
4. Abuse of alcohol, narcotics or drugs
5. Pregnancy, breastfeeding or current pregnancy wish. Fertile women must use effective anticonception, (hormonal contraception, contraceptive injection, implant or patches, intrauterine system and device, vaginal ring).
6. Treatment with all pain modulating drugs, e.g. all analgesics, antidepressants, antiepileptica and other types of medication with pain relieving properties must be discontinued at least two weeks before the treatment phase.
7. Imipramine treatment in sufficient dosage within the last year, i.e. 25 mg daily continuously for at least 8 weeks.
8. Allergy to study medication or excipients in study medication.
9. Patients with previous med myocardial infarction, congestive heart failure, signs of conduction defects or abnormalities on ECG (first degree AV-block, bundle branch block or prolonged QT-interval), narrow-angle glaucoma, porphyria, inherited galactose intolerance, epilepsy, hepatic insufficiency and severe renal impairment
10. Simultaneous use of:

    * antipsychotics
    * oral anticoagulants
    * diuretics
    * sympathomimetics and CNS-stimulating drugs (amphetamine-like drugs)
    * all serotonergic drugs, e.g. SSRI, SNRI and TCA, the dietary supplement hypericum perforatum, non-selective, irreversible or selective, reversible monoamine oxidase (MAO) inhibitors, triptans, tramadol, pethidin and tryptophan
    * the drugs cimetidine (H2-antagonist), quinidine (antiarrythmics), clonidine (antihypertensive), fluconazol (antimycotics), clindamycin, clarithromycin, erythromycin (antibiotics), droperidol (anaesthetic), levodopa (antiparkinson), mefloquine (antimalaria), phenytoin, barbiturates, carbamazepin (antiepileptica)
    * Bupropion (tobacco dependence), celecoxib (NSAID), cinacalcet (antiparathyroid drug), duloxetine (SNRI), flufenazin (antipsychotic), fluoxetin (SSRI), gefitinib (antineoplastic), moclobemid (MAO), paroxetine, Sertraline (SSRI), Terbinafine (antimycotics), Yohimbin (erectile dysfunction) samt fluvoxamin (SSRI), ciprofloxacin and enoxacin (microbiotic), because plasma concentration of Imipramine can increase with the simultaneous use of these potent CYP2D6- and CYP1A2- inhibitors

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Global Clinical Improvement Scale | After 13 weeks
  Questionnaire, patient-rated improvement of health since the beginning of the study.

SECONDARY OUTCOMES:
SF-36 | At 1 and 13 weeks
  Questionnaire, patient-rated. Assessment of physical, social and mental functioning
Visual Analogue Scale for pain and worst symptom | At 1 and 13 weeks
Symptom Checklist (SCL) | At 1, 3 and 13 weeks
Functional Illness Checklist (FIC) | At 1, 3 and 13 weeks
WHODAS II | At 1 and 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Per k Fink, dr.med, Principal Investigator — Aarhus University Hospital
Locations (1):
- Research Clinic for Functional Disorders, Aarhus, Denmark

REFERENCES:
- [Result] Agger JL, Schroder A, Gormsen LK, Jensen JS, Jensen TS, Fink PK. Imipramine versus placebo for multiple functional somatic syndromes (STreSS-3): a double-blind, randomised study. Lancet Psychiatry. 2017 May;4(5):378-388. doi: 10.1016/S2215-0366(17)30126-8. Epub 2017 Apr 10. PMID 28408193